CLINICAL TRIAL: NCT06782269
Title: Incidence of Subtalar Joint Fusion After Isolated Ankle Fusion
Status: Not yet recruiting | Type: Observational
Sponsor: Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: RL1901
Record Dates: First submitted 2024-09-05; First posted 2025-01-17 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Ankle Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ankle fusion — fusion of ankle joint

SUMMARY:
It is important to know a truer incidence of the need for subtalar and midfoot fusions, following an isolated ankle fusion, in order to better inform our patients of the likelihood of needing further surgery in the future. It is also important to understand whether pre-existing radiological arthrosis is likely to lead to the need for a fusion in the future and also how important the alignment of the ankle joint, after a fusion, may influence that.

The aim of the study is to review the patients' notes and radiology who have had a previous isolated ankle fusion and then to see whether they subsequently required further surgery.

DETAILED DESCRIPTION:
Isolated ankle fusion is normally regarded as a good operation producing good pain relief and allowing patients to function well. Patients will have an early heel rise when walking and although that is often not immediately perceptible to an onlooker, it does increase the stress on the neighbouring subtalar and Chopart joints. Radiologically, subtalar joint arthrosis is common following isolated ankle fusions but not necessarily clinically symptomatic. The long term incidence of subsequent ipsilateral subtalar or Chopart joint fusions is not well known. Various different studies have shown a prevalence of osteoarthrosis (radiologically) of 24-100% in the subtalar joint and reported 84% of patients complaining of pain after 10 years. The prevalence in the Chopart joints has been reported to vary between 18-77%.

This is an observational study reviewing medical records and radiology of patients who have had an isolated ankle fusion. The data will be analysed using basic statistics with logistic regression modelling.

ELIGIBILITY:
Inclusion Criteria:

Any patient who has had an isolated ankle fusion and is over the age of 18 years old.

Exclusion Criteria:

Participants younger than 18 years old.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had an isolated ankle fusion.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of subtalar and midfoot fusions after isolated fusion of the ankle joint | A retrospective data collection following patients from surgery to now.
  To look at the incidence of subtalar and midfoot fusions after an isolated ankle fusion and what factors influenced this.

IPD SHARING:
Plan to Share IPD: No